CLINICAL TRIAL: NCT01767168
Title: Trial of Diagnostic Accuracy for the Prediction of Persistent Postoperative Pain After Breast Cancer Surgery Using a Conditioned Pain Modulation Test
Brief Title: Study to Test the Value of a Pain Modulation Test in Predicting Persistent Postoperative Pain After Breast Cancer Surgery
Acronym: PREDO
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Benno Rehberg-Klug, médecin adjoint agrégé, University Hospital, Geneva
Other Study IDs: CER 10-218; matped 10-054 (Other: local ethics committee)
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Pain; Acute Pain
MeSH Terms: conditions — Chronic Pain; Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — venous blood sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: comprehensive preoperative testing for risk factors of persistent postoperative pain — nociceptive reflex threshold, pain threshold, CPM-effect of hot water bath, pain sensitivity questionnaire, STAI, BDI, fear of surgical consequences

SUMMARY:
The purpose of this study is to test the hypothesis that a preoperative test of pain modulation predicts persistent pain 4 months after breast cancer surgery. In addition, a risk score for the prediction of persistent pain will be developed from parameters available before surgery.

ELIGIBILITY:
Inclusion Criteria:

* age >=18 years
* American Society of Anesthesiology functional status I-III
* able to read and understand the information sheet and give informed consent

Exclusion Criteria:

none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women scheduled for any type of breast cancer surgery in a university hospital breast cancer center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-05; Primary Completion 2015-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
prevalence of pain at the site of surgery | 4 months postop
  clinically important pain defined as either necessitating analgesic treatment or having an intensity of more than 3/10 at rest or 5/10 on movement, at 4 months after surgery

SECONDARY OUTCOMES:
acute pain | 24h
  maximum pain >3/10
subacute pain | 1 week
  average pain, maximum pain >2
prevalence of pain necessitating analgesics at the site of surgery | 4 months
prevalence of pain at the site of surgery | 8 months
prevalence of pain at the site of surgery | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Benno Rehberg-Klug, MD, Principal Investigator — Dept of Anesthesiology, HUG
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva, Switzerland